CLINICAL TRIAL: NCT04915157
Title: Efficacy of Spinal Cord Stimulation in Patients With Refractory Angina Pectoris; a Randomized Controlled Trial
Brief Title: Efficacy of Spinal Cord Stimulation in Patients With Refractory Angina Pectoris
Acronym: SCRAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Inge Wijnbergen, Principal Investigator, Catharina Ziekenhuis Eindhoven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCRAP
Record Dates: First submitted 2021-05-11; First posted 2021-06-07 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Refractory Angina Pectoris; Spinal Cord Stimulation
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 fashion to either Group A (High Density stimulation - No stimulation) or Group B (No stimulation - High Density stimulation).
  All patients will receive an implanted spinal cord stimulator.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One nurse will perform the randomization and know to which group the patient was randomized. The same nurse will input the correct settings into the spinal cord stimulator. The other investigators, the participant, care provider and outcomes assessor will remain masked during the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: High Density stimulation - No Stimulation (Other): Patients in this group will receive high density stimulation (parasthesia free form of stimulation) during the first 6 months of the study period. After 6 months cross-over will take place and patients will receive no stimulation during the final 6 months of the study period.
  Interventions: Device: Spinal Cord Stimulator
- Group B: No Stimulation - High Density Stimulation (Other): Patients in this group will receive no stimulation during the first 6 months of the study period. After 6 months cross-over will take place and patients will receive high density stimulation (parasthesia free form of stimulation) during the final 6 months of the study period.
  Interventions: Device: Spinal Cord Stimulator

INTERVENTIONS:
Device: Spinal Cord Stimulator — All patients will receive an implanted spinal cord stimulator.
  Other Names: Medtronic PrimeADVANCED™ SureScan® myStim & Vectris Compact™ SureScan MRI electrode

SUMMARY:
There are a growing number of patients with refractory angina pectoris (RAP). RAP is defined as a 'chronic condition (> three months) characterized by diffuse coronary artery disease in the presence of proven ischemia, which is not amendable to a combination of medical therapy, angioplasty or coronary bypass surgery'. These patients are severely restricted in performing daily activities due to debilitating angina complaints, leading to a decreased quality of life.

Spinal cord stimulation (SCS) is a last resort treatment option for patients with RAP. SCS is a device with a lead located in the thoracic epidural space and an Implantable Pulse Generator (IPG) in the abdomen or buttock that provides neurostimulation. Four possible mechanisms explaining the beneficial effects of SCS on RAP have been described: reduction of pain perception, decreased sympathetic tone, reduced myocardial oxygen demand, and improved coronary microcirculatory blood flow.

Research into the effect of SCS on RAP up to date have mainly been observational studies, with only four placebo-controlled randomized controlled trials. All studies confirm that treatment with SCS leads to a reduction in the number of angina pectoris attacks. What is currently not clear, is whether there is a placebo effect as results vary between the studies. One study looked at the effect of SCS in patients with RAP on the reduction of ischemia (using MIBI-SPECT) with no control arm. After 12 months myocardial ischemia was reduced, but not after three months of treatment. Leading to the conclusion that the reduction is myocardial ischemia was not a direct effect of SCS, but rather due to better coronary collateralization.

The 2020 ESC guideline 'chronic coronary syndromes' mentions non-existing to promising levels of evidence with regard to treatment options in patients with RAP and concludes that SCS may be considered (Class IIB; level of evidence B). It concludes that 'larger RCTs are required to define the role of each treatment modality for specific subgroups, to decrease non-responder rates and ascertain benefit beyond potential placebo effects'.

The aim of the current randomized controlled trial (double-blind, cross-over, placebo-controlled, single center) is to determine if high density spinal cord stimulation, a paresthesia free form of stimulation, leads to a significant reduction in myocardial ischemia (using PET with Rubidium-82 as tracer) in patients with refractory angina pectoris.

All patients included in this study will receive an implanted spinal cord stimulator after a positive TENS treadmill outcome and proven ischemia using the imaging modality PET with Rubidium-82 as tracer. Using a cross-over design all patients will have a 6 month period with high density stimulation and 6 month period of no stimulation. Randomization will determine in which order the patient receives these treatments. Both the patient and the treating physicians are blinded for this randomization process. At baseline a 6-minute walking test, the Seattle Angina Questionnaire, the RAND-36 questionnaire, the NRS scale and the CCS class will be performed/filled out.

Cross-over takes place at 6 months (switch from high density stimulation to no stimulation or vice versa) prior to which the PET scan is repeated, as well as the 6-minute walking test, the Seattle Angina Questionnaire, the RAND-36 questionnaire, the NRS-scale and the CCS-class.

At the end of the study period (12 months) the PET scan is repeated, as well as the 6-minute walking test, the Seattle Angina Questionnaire, the RAND-36 questionnaire, the NRS-scale and the CCS-class.

ELIGIBILITY:
Inclusion Criteria:

* Refractory Angina Pectoris:

  * Stable angina pectoris CCS class III or IV, with a minimum of 5 episodes of angina pectoris over the course of one week, during a minimum period of three months prior to screening
  * Coronary angiogram (CAG) performed within the last 12 months showing significant coronary artery disease defined as at least one coronary artery stenosis of >75% or 50 - 75% with proven ischaemia (see below), not suitable for revascularisation. Confirmed by one (or two in case of doubt) interventional cardiologist based on CAG images.
  * Optimal anti-anginal medication. Patients should at least use the maximal tolerable dose of a b-blocker, calcium channel blocker and short- and/or long-acting nitrate. If the patient doesn't use one of these groups of medication the reason (side-effects) should be clear.
* Proven ischemia:

  * MIBI-SPECT: summed stress score (SSS) of at least 1, in combination with summed difference score (SDS) of at least 1 (1-4 mild ischaemia, > 4 moderate to severe ischaemia).
  * FFR: < 0.80, with no intervention options (determined by interventional cardiologist)
  * MRI perfusion: ≥ 1 segment of subendocardial hypoperfusion during stress perfusion, not present at rest and no matching fibrosis (using 16 segment AHA heart model)
  * PET: Semi-quantitative measurement: SSS score of at least 1, in combination with SDS score of at least 1 (1-4 mild ischaemia, > 4 moderate to severe ischaemia). Quantitative measurement: reduced myocardial perfusion reserve.
* No revascularisation (PCI and/or CABG) performed between ischaemia testing and study inclusion.
* Age > 18 years

Exclusion Criteria:

* Acute coronary syndrome (ACS) during the three month period prior to screening
* Life expectancy less than 12 months
* Inability to perform a 6-minute walking test
* Inability to give informed consent
* No proven ischemia
* Spinal cord disease which could prevent correct positioning of the lead in the epidural space; to be determined by the anaesthesiologist performing the implantation
* Anticoagulation therapy that cannot be stopped/bridged prior to spinal cord stimulator implantation
* Inadequate paraesthesia coverage, during implantation, of the thoracic region where angina complaints are localized
* Pregnancy
* Mild Cognitive Impairment or dementia
* Concomitant symptomatic valvular heart disease including severe aortic stenosis and/or regurgitation, severe mitral valve stenosis and/or regurgitation or severe tricuspid valve regurgitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Myocardial ischaemia | 6 months
  The primary endpoint is the change in the percentage of myocardial ischaemia (% of left ventricular myocardium) measured using PET perfusion scan at the end of the six month period of HD stimulation compared to baseline.

SECONDARY OUTCOMES:
Patient condition | From date of randomization until six and twelve months later
  Patient condition measured using the 6-minute walking test
Frequency of angina pectoris attacks | From date of randomization until six and twelve months later
  Frequency of angina pectoris attacks measured using the Seattle Angina Questionnaire; scale 0 - 100 with higher scores representing a better outcome.
Severity of angina pectoris attacks | From date of randomization until six and twelve months later
  Severity of angina pectoris attacks using the Numeric Rating Scale (NRS-scale); scale 0 - 10 with higher scores representing a worse outcome.
Grading of angina pectoris | From date of randomization until six and twelve months later
  Grading of angina pectoris using the Canadian Cardiovascular Society (CCS) class; grading scale of I - IV with higher scores representing worse outcome.
Frequency of short-acting nitroglycerin use | From date of randomization until six and twelve months later
  Frequency of short-acting nitroglycerin use measured using the Seattle Angina Questionnaire; scale 0 - 100 with higher scores representing a better outcome.
Quality of life outcome | From date of randomization until six and twelve months later
  Quality of life outcome measured using the RAND 36-Item Health Survery (RAND-36 questionnaire); scale 0 - 100 with higher scores representing a better outcome.
Hospital admissions due to acute coronary syndrome | From date of randomization until six and twelve months later
  Number of hospital admissions due to acute coronary syndrome (ACS)
Revascularization | From date of randomization until six and twelve months later
  Occurence of revascularization (CABG and/or PCI)
Emergency room visits due to angina pectoris | From date of randomization until six and twelve months later
  Number of presentations at the emergency room due to angina pectoris
Cardiovascular mortality | From date of randomization until six and twelve months later
  Occurence of cardiovascular mortality
Changes in regional and global myocardial blood flow and myocardial flow reserve | From date of randomization until six and twelve months later
  Changes in the regional and global myocardial blood flow and myocardial flow reserve measured using PET perfusion scan

OTHER OUTCOMES:
Device infection | From date of randomization until six and twelve months later
  Number of device infections (lead and/or battery)
Device dislocation | From date of randomization until six and twelve months later
  Number of device dislocations (lead and/or battery)
Lead fractures | From date of randomization until six and twelve months later
  Number of lead fractures/breakages
Lead failure | From date of randomization until six and twelve months later
  Number of lead failures
Battery End of Life (EOL) | From date of randomization until six and twelve months later
  Number of battery End of Life (EOL)

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Vervaat FE, van der Gaag A, Smetsers C, Barneveld PC, Van't Veer M, Teeuwen K, van Suijlekom H, Dekker L, Wijnbergen IF. Design and rationale of the efficacy of spinal cord stimulation in patients with refractory angina pectoris (SCRAP) trial. Clin Cardiol. 2023 Jun;46(6):689-697. doi: 10.1002/clc.24016. Epub 2023 Apr 4. PMID 37013654